CLINICAL TRIAL: NCT05814185
Title: The Effect of Two and Four Activations Per Day of the Periodontal Distractor on Pain Intensity and Pulp Vitality of Maxillary Canine: Randomized Clinical Trial
Brief Title: Distractor Effect on Pain and Vitality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Alaa Mossad, Assistant lecturer of orthodontics, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDL distractor
Record Dates: First submitted 2023-02-27; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Distraction of Bone
MeSH Terms: conditions — Diastasis, Bone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Canine retraction was done by periodontal distractor with two activations per day. (Experimental): group 1
  Interventions: Device: Periodontal distractor
- Canine retraction was done by periodontal distractor with four activations per day. (Experimental): group 2
  Interventions: Device: Periodontal distractor

INTERVENTIONS:
Device: Periodontal distractor — different activation protocols of periodontal distractor

SUMMARY:
The aim of the present study was to evaluate the effect of two and four activations /day of periodontal distractor on pain intensity and pulp vitality of maxillary canine.

DETAILED DESCRIPTION:
Orthodontic therapy is generally referred to as a lengthy process because a good orthodontic treatment normally takes 18 to 24 months to finish.

Long-term orthodontic treatment has a number of disadvantages, including as poor psychosocial effects on patients, white spots, long-term enamel damage, gingival recession, and root resorption.

The rate of tooth movement that can be achieved is a major determinant of orthodontic treatment time. Many studies have been conducted to determine the pace of orthodontic tooth movement. The majority of these studies demonstrate about 1mm of tooth movement per month.

As a result, finding treatment options that reduce treatment time without compromising results is a main focus of orthodontic research.

The approaches for hastening tooth movement rely on inducing a biological tissue reaction. These procedures are classified into two types based on their level of intrusion: conservative (biological, physical, and biomechanical measures) and surgical techniques Prostaglandins are the most often used biological agents , interleukins , leukotriene , vitamin D platelet rich plasma .Mechanical or physical approach include direct electrical current , pulsed electromagnetic field , low-energy laser , and Vibration Oral surgical procedures quicken orthodontic treatment by affecting the continuity of the alveolar bone resulting in a decrease in bone density and a corresponding reduction in the bone's resistance to orthodontic tooth movement . Surgical approach depends on Regional Acceleratory Phenomenon (RAP) which is a method to speed up orthodontic treatment by accelerating bone remodeling rates and bone density. The RAP is a series of tissue reactions that occur as a damaged bone heals . These surgical methods including corticotomy , bone perforation , Distraction osteogenesis is also one of surgical methods that allow rapid canine retraction .

The technique of distraction of the periodontal ligament (PDD) was introduced for rapid tooth movement then, dento alveolar distraction (DAD) was performed to achieve rapid tooth movement using the principles of distraction osteogenesis The canine was distracted by distractor twice daily for a total about 0.4 mm per day . It has been reported in literature that up to 2 mm is distracted per day (four activations of 0.5 mm each) . The distractor was activated till the distal surface of canine became in contact with the mesial surface of second premolar.

Previous Studies of periodontal distractor have been mainly focused on the assessment of the rate and angular changes on retracted canine. No clinical study has attempted to investigate pain intensity or pulp vitality for both activation protocols of periodontal distractor during rapid canine retraction. Therefore, the aim of the present study was to evaluate the effect of two and four activations/day of periodontal distractor on pain intensity and pulp vitality of maxillary canine.

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic Patients need extraction of first permanent premolar for orthodontic reasons (dentoalveolar maxillary protrusion, Class II div 1 malocclusion)
* No history of previous orthodontic treatment
* Absence of any systemic disease
* Good oral hygiene and healthy gums look, with no signs of redness, edema, or bleeding during brushing (periodontal inflammation)
* Highly motivation and cooperation

Exclusion Criteria:

* Medically compromised patients
* Use of medication that may affect tooth movement during the period of the study

Ages: 16 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
pain intensity | 1st 48 hour after intervention (from the time of distractor placement until the end of the 2nd day)
  evaluation of pain intensity by Visual Analogue scale.minimum 0 and maximum value 10.
pain intensity | during each activation of the distractor,(up to 1 minute during moving the key of distractor)
  evaluation of pain intensity by Visual Analogue scale.minimum 0 and maximum value 10
pain intensity | up to 6 hours on the four activations group and up to 12 hours on two activations group.
  evaluation of pain intensity by Visual Analogue scale. minimum 0 and maximum value 10
pulp vitality | before and after canine retraction (up to one month)
  vitality by Electric pulp tester.positive reading is better

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M. Eldriny, Lecturer, Principal Investigator — Assistant Lecturer of Orthodontics,Al Azhar University, Cairo, Egypt.; Ahmed A. Salama, professor, Study Director — Professor of Orthodontics, Al Azhar University, Cairo, Egypt.; Osama S. El-Shal, professor, Study Director — Professor of periodontology Al Azhar University, Cairo, Egypt.; Maha M. Mohamed, professor, Study Director — Assistant professor of Orthodontics, Al Azhar University, Cairo, Egypt.
Locations (1):
- Faculty of Dental Medicine, for Girls, Al Azhar University, Cairo, Nasr City, Egypt

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-10-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT05814185/Prot_SAP_ICF_000.pdf